CLINICAL TRIAL: NCT03036579
Title: Clinical Evaluation of Chairside Computer Assisted Design/Computer Assisted Machining (CAD/CAM) Zirconia-reinforced Lithium Silicate Ceramic Crowns
Brief Title: Celtra Duo Computer Assisted Design/Computer Assisted Machining (CAD/CAM) Dental Crown Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID, loss of funding
Sponsor: University of Michigan (Other)
Collaborators: Dentsply Sirona Inc. (Industry)
Responsible Party: Principal Investigator, Dennis J. Fasbinder, DDS, Clinical Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00103921
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Results first posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Fractured Tooth; Decayed Tooth; Unsatisfactory Restoration of Tooth
Keywords: CAD/CAM; Ceramic; Crown
MeSH Terms: conditions — Tooth Fractures

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Final surface fabrication was not identified in the treatment process until the crown was milled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Glazed Fired, Calibra Céram (Experimental): Celtra Duo crowns will be glaze-fired in a porcelain oven and cemented with Calibra Ceram Cement
  Interventions: Device: Celtra Duo
- Hand Polished, Calibra Universal (Experimental): Celtra Duo crowns will be hand-polished and cemented with Calibra Universal Cement
  Interventions: Device: Celtra Duo

INTERVENTIONS:
Device: Celtra Duo — Full ceramic crowns will be made from the high strength ceramic, Celtra Duo.

SUMMARY:
This investigation will be a clinical trial to study the performance of a newly developed high strength ceramic material for crowns. The ceramic has been approved by the FDA for patient treatment. A computer technique will be used to fabricate the crowns in a single appointment without the need for a temporary crown or second appointment. Two adhesive resin cement techniques will be used to hold the crown to the tooth and they will be evaluated for creating sensitivity to the tooth. The purpose of the study is to measure how well the high strength crowns function over an extended period of time.

DETAILED DESCRIPTION:
The study will be composed of two groups of 50 crowns placed in adult patients that have been identified as requiring at least one crown on a posterior tooth. A maximum of two crowns per patient will be completed. All the crowns will be made from the same high strength ceramic material (Celtra Duo/Dentsply Sirona). The two groups of crowns will be made using two different processes to create the surface texture and finish for the crown. One group of Celtra Duo crowns (Group 1) will be glaze-fired in a porcelain oven and the second group (Group 2) will be hand-polished. All the crowns will be cemented using two adhesive techniques. All of the oven-fired, glazed crowns will be cemented using the self-etching, self-adhesive resin cement technique (Calibra Universal Cement/Dentsply). All of the hand polished crowns will be cemented using an adhesive bonding technique using Prime & Bond Elect (Dentsply) with a dual cured resin cement (Calibra Ceram/Dentsply). The crowns are planned to be evaluated at 6 months, 1 year, 2 years, 3 years, and if funding permits, 4 years, and 5 years. At each appointment an examination of the crown will be completed as well as clinical photographs, an intraoral digital scan, and impression of the crown.

ELIGIBILITY:
Inclusion Criteria:

* must have at least one carious lesion or defective restoration or fractured tooth in a molar or premolar
* reason for restoration should extend more than one-half the intercuspal width of the tooth requiring a full crown restoration
* Teeth to be vital and asymptomatic prior to treatment
* No more than two restorations will be placed per patient. If a patient presents with more than two acceptable teeth for the study, molar teeth will be included prior to premolar teeth.

Exclusion Criteria:

* Devital or sensitive teeth
* Teeth with prior endodontic treatment of any kind
* Teeth with a history of direct or indirect pulp capping procedures
* Patients with significant untreated dental disease to include periodontitis and rampant caries
* Pregnant or lactating women
* Patients with a history of allergies to any of the materials to be used in the study
* Patients unable to return for the recall appointments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2015-11; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis J Fasbinder, DDS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Recall at 5 years not funded by sponsor, therefore data not collected up to 5 years
Units Other Than Participants: tooth
Period: Baseline
Arm/Group | Glazed Fired, Calibra Céram | Hand Polished, Calibra Universal
Started | 41; 50 tooth (some participants had 2 teeth restored with crowns) | 32; 50 tooth (some participants had two teeth restored with crowns)
Completed | 41; 50 tooth | 32; 50 tooth
Not Completed | 0; 0 tooth | 0; 0 tooth
Period: 6 Months
Arm/Group | Glazed Fired, Calibra Céram | Hand Polished, Calibra Universal
Started | 41; 50 tooth | 32; 50 tooth
Completed | 41; 50 tooth | 32; 50 tooth
Not Completed | 0; 0 tooth | 0; 0 tooth
Period: 1 Year
Arm/Group | Glazed Fired, Calibra Céram | Hand Polished, Calibra Universal
Started | 41; 50 tooth | 32; 50 tooth
Completed | 41; 50 tooth | 32; 50 tooth
Not Completed | 0; 0 tooth | 0; 0 tooth
Period: 2 Years
Arm/Group | Glazed Fired, Calibra Céram | Hand Polished, Calibra Universal
Started | 41; 50 tooth | 32; 50 tooth
Completed | 40; 49 tooth | 32; 50 tooth
Not Completed | 1; 1 tooth | 0; 0 tooth
Not completed — Lost to Follow-up | 1 | 0
Period: 3 Years
Arm/Group | Glazed Fired, Calibra Céram | Hand Polished, Calibra Universal
Started | 41; 50 tooth (The participant lost to follow up in year 2 participated in year 3 which is why the number of participants to start in year 3 does not equal those who completed year 2.) | 32; 50 tooth
Completed | 41; 50 tooth | 31; 49 tooth
Not Completed | 0; 0 tooth | 1; 1 tooth
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Number of teeth restored with crowns
Units Other Than Participants: number of teeth restored with crowns
Groups:
- Total: Total of all reporting groups
Arm/Group | Glazed Fired, Calibra Céram | Hand Polished, Calibra Universal | Total
Number analyzed (Participants) | 41 | 32 | 73
Number analyzed (number of teeth restored with crowns) | 50 | 50 | 100
Age, Customized [Count of Participants; unit: Participants] — Age data not collected from any participant Population: Age data not collected from any participant
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 23 | 49
  Male | 15 | 9 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Crown Failure
Description: Crown failure includes fracture of the crown or loss of the crown requiring placement of a new crown at any time between delivery and three years.
Time Frame: from delivery of the crown up to 3 years
Population: teeth restored with crowns
Measure: Number; unit: crowns
Units Other Than Participants: Teeth
Arm/Group | Glazed Fired, Calibra Céram | Hand Polished, Calibra Universal
Number analyzed (Participants) | 41 | 32
Number analyzed (Teeth) | 50 | 50
crowns | 5 | 5

2. Secondary Outcome: Crown Loss of Retention
Description: Loss of retention is measured as detachment of the crown from the tooth without fracture of the crown requiring recementation of the crown.
Time Frame: 3 years
Population: number of crowns
Measure: Number; unit: crowns
Units Other Than Participants: Teeth
Arm/Group | Glazed Fired, Calibra Céram | Hand Polished, Calibra Universal
Number analyzed (Participants) | 41 | 32
Number analyzed (Teeth) | 50 | 50
crowns | 2 | 0

3. Secondary Outcome: Tooth Sensitivity
Description: Tooth Sensitivity is evaluated as either "0" if the subject reports that there is NO sensitivity for the tooth with the study crown, or "1" if the subject reports that there IS tooth sensitivity to hot/cold or biting pressure. The better outcome is to have NO tooth sensitivity. The number of teeth with tooth sensitivity are listed below.
Time Frame: 3 years
Population: number of teeth with crown
Measure: Number; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | Glazed Fired, Calibra Céram | Hand Polished, Calibra Universal
Number analyzed (Participants) | 41 | 32
Number analyzed (Teeth) | 50 | 50
Teeth | 0 | 0

4. Secondary Outcome: Margin Staining
Description: Margin Staining is evaluated as either "0" if there is NO staining at the crown margin where it meets the tooth, or "1" if there IS staining at the crown margin where it meets the tooth. The better outcome is to have NO margin staining. The number of teeth with margin staining are listed below.
Time Frame: from delivery of the crown up to 3 years
Population: number of crowns
Measure: Number; unit: crowns
Units Other Than Participants: Teeth
Arm/Group | Glazed Fired, Calibra Céram | Hand Polished, Calibra Universal
Number analyzed (Participants) | 41 | 32
Number analyzed (Teeth) | 50 | 50
crowns | 2 | 2

ADVERSE EVENTS:
Time Frame: from baseline to 3 years
Arm/Group | Glazed Fired, Calibra Céram | Hand Polished, Calibra Universal
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/32
Other Adverse Events (participants affected / at risk) | 0/41 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-19): https://cdn.clinicaltrials.gov/large-docs/79/NCT03036579/Prot_SAP_000.pdf